CLINICAL TRIAL: NCT03662373
Title: Sperimentazione Clinica Del Sistema INSIDE - Innovative SolutIons for DosimEtry in Hadrontherapy - Per il Monitoraggio Del Trattamento in Adroterapia
Brief Title: Innovative SolutIons for DosimEtry in Hadrontherapy (INSIDE)
Acronym: INSIDE
Status: Recruiting | Type: Observational
Sponsor: CNAO National Center of Oncological Hadrontherapy (Other)
Responsible Party: Sponsor
Other Study IDs: CNAO-OSSINSIDE-02-18
Record Dates: First submitted 2018-07-03; First posted 2018-09-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-02

CONDITIONS: Particle Therapy
Keywords: on line monitoring; PET in beam; Hadrontherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- carbon ions radiation therapy: the group of patients treated with carbon ion radiation therapy, affected by one of the four pathologies foreseen in inclusion criteria
  Interventions: Radiation: carbon ions radiation therapy
- protons radiation therapy: the group of patients treated with proton radiation therapy, affected by one of the four pathologies foreseen in inclusion criteria
  Interventions: Radiation: protons radiation therapy

INTERVENTIONS:
Radiation: carbon ions radiation therapy — Carbon ion radiation therapy to treat adenoid cystic carcinoma, skull base (clivus) chordoma.
  Other Names: particle therapy
  Groups: carbon ions radiation therapy
Radiation: protons radiation therapy — Proton radiation therapy used to treat meningioma and squamocellular rhinopharynx carcinoma
  Other Names: particle therapy
  Groups: protons radiation therapy

SUMMARY:
The study aim is to test the clinical feasibility and effectiveness of an online qualitative monitoring device named INSIDE system during hadrontherapy treatments.

This instrumentation is composed by detectors able to acquire secondary signals generated by the interaction of the primary beam with human tissues. From these measurements performed during irradiation, the INSIDE system estimates the particle beam range inside the patient's body and check the compliance of the ongoing treatment with the clinical prescription, with the aim to optimize the delivered dose.

The study aims to longitudinally monitor patients treated with hadrontherapy at the Italian National Centre of Oncological Hadrontherapy (CNAO) in Pavia in order to:

* evaluate the stability of the INSIDE system response and the significance of the monitoring measurement;
* study the clinical tolerances between ongoing and prescribed treatments within which the differences in particle range are not clinically relevant;
* assess what impact an instrument such as the INSIDE system can have on the clinical routine;
* evaluate the benefits of such a monitoring system with respect to treatment planning constraints.

DETAILED DESCRIPTION:
A treatment monitoring instrumentation is highly demanded to maximize the benefits of hadrontherapy from the increased conformation of the released dose to the tumor volume with respect to the conventional radiotherapy.

Since almost all the energy of the charged particles is deposited in the end of their track (Bragg Peak region), the verification of the particle range by experimental measurements, performed during treatment delivery, can help to increase the therapy effectiveness while better sparing healthy tissues.

The INSIDE system is an innovative bi-modal instrumentation consisting of an in-beam Positron Emission Tomography (PET) scanner, to detect annihilation photons coming from positron isotope emitters, and a Dose Profiler to collect signals from charged particles emitted during treatment (e.g. protons in the case of carbon ion treatments).

The in-beam PET scanner is composed by two opposite panels of detectors placed above and below the patient bed, respectively. The Dose Profiler is positioned above the patient with an angle of 60°, forwardly with respect to the beam direction.

The INSIDE system is a passive instrumentation, i.e. no additional dose has to be released to the patient for particle range verification.

The INSIDE detectors are mounted on a mobile support and, immediately before the treatment delivery, they will be placed around the patient in the acquisition position, thanks to a dedicated hooking system designed to guarantee the maximum precision and accuracy in the particle range verification.

The INSIDE system mechanics is compatible with multi fields irradiation of patients affected by pathologies of Head-and-Neck and Brain districts.

In the clinical trial, patients affected by four selected pathologies will be included: meningioma and nasopharynx cancers treated with proton beams, Adenoid Cystic Carcinoma (ACC) and clival chordoma treated with carbon ion beams. These were chosen in order to study both projectile particles available at the CNAO centre (i.e., protons and carbon ions), and target specific pathologies which should most benefit from the range monitoring provided by the INSIDE system. Among them are cancers for which an early response is commonly observed and tumors which are located near cavities that can be filled with either water-like material (such as cancerous mass and inflamed tissues) or air.

The patients will undergo a longitudinal protocol of measurements in order to verify the agreement between the ongoing treatment and the prescription throughout the complete treatment period (lasting in average about 4-6 weeks for the selected pathologies).

ELIGIBILITY:
Inclusion Criteria:

* patients treated at CNAO with protons or carbon ions with horizontal beam line.
* meningioma, ACC, skull base (clivus) chordoma, squamous cellular rhinopharynx carcinoma
* full compatibility of the INSIDE monitoring system with all beam delivery devices in the established irradiating position
* all emergency procedures are possible notwithstanding INSIDE system positioned.
* signed written informed consent by patient.

Exclusion Criteria

* missing informed consent
* not affected by one of the selected pathologies
* failure of pre-treatment compatibility technical assessment
* failure of pre-treatment emergency procedures check
* medical or individual reasons (i.e. short time test needed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is represented by all patients undergoing to treatment at CNAO, selected on the pathology and on the particle used for their radiation therapy. 40 patients affected by one of the four pathologies foreseen and which can offer morphological variations during treatment cycle.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
particles ranges | average of 5 weeks (as a treatment duration)
  evaluate the quality of treatments in term of data collection and of particles range evaluated with PET scanner and Monte Carlo simulations
particles ranges for each pathology considered | 4 months
  statistical analysis to assess the evaluations of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Viviana Vitolo, MD, Principal Investigator — CNAO National Center of Oncological Hadrontherapy
Locations (1):
- CNAO, Pavia, Pavia, Italy